CLINICAL TRIAL: NCT03014843
Title: The Effect of Naloxone and Mehtylnaltrexone on Esophageal Sensitivity in Healthy Volunteers: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Effect of Naloxone and Methylnaltrexone on Esophageal Sensitivity in Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: S54661
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Endogenous and Esophageal Sensitivity
Keywords: Esophagal sensitivity, GERD, endogenous opiods
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Naloxone; methylnaltrexone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naloxone (Active Comparator): Administration of a centrally acting µ-opioid receptor antagonist Naloxone (20µg/kg/h intravenous infusion after 0.4mg bolus) to investigate the effect of esophageal sensitivity assessed by multimodal esophageal stimulation.
  Interventions: Drug: Naloxone
- Methylnaltrexone bromide (Active Comparator): Administration of a peripherally acting µ-opioid receptor antagonist Methylnaltrexone (12mg/0.6mL subcutaneous injection) to investigate the effect of esophageal sensitivity assessed by multimodal esophageal stimulation.
  Interventions: Drug: Methylnaltrexone Bromide
- Placebo (Placebo Comparator): Administration of placebo injection (1mL 0.9% saline IV or 0.6 IM) as a control condition to compare to the administration of naloxone or methylnaltrexone bromide in the multimodal esophageal stimulation protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naloxone — 20µg/kg/h intravenous infusion after 0.4mg bolus of Naloxone and 0.6mL IM NaCl (0.9%) injection (this step is necessary to keep the subject blinded for the condition since nalaxone and methylnaltrexone have different administration routes)
  Other Names: Naloxon, B.Braun
  Arms: Naloxone
Drug: Methylnaltrexone Bromide — 12mg/0.6mL subcutaneous injection and 1mL bolus of NaCl (0.9%) followed by intravenous infusion (this step is necessary to keep the subject blinded for the condition since nalaxone and methylnaltrexone have different administration routes)
  Other Names: Relistor
  Arms: Methylnaltrexone bromide
Other: Placebo — 0.6 mL of NaCl 0.9% will be injected IM and 1mL bolus injection of NaCl(0.9%) will be administered IV followed by IV NaCl 0.9% infusion
  Other Names: Saline solution (0.9% NaCl)
  Arms: Placebo

SUMMARY:
The aim of this study was to investigate the effect of naloxone (IV or IM administration) and methylnaltrexone (subcutaneous administration) on esophageal sensitivity, in a group of healthy volunteers in order to evaluate the role of endogenous opiods in symptom perception in gastro-esophageal reflux disease. Esophageal sensitivity was assessed by using a multimodal esophageal stimulation protocol where sensitivity to thermal, mechanical, electrical and chemical stimulation was tested.

DETAILED DESCRIPTION:
INTRODUCTION Gastroesophageal reflux disease (GERD), defined as the presence of symptoms or lesions that can be attributed to the reflux of gastric contents into the esophagus, is an increasingly prevalent condition in Western societies. The most typical symptoms are heartburn and regurgitation, but GERD can manifest itself through a variety of esophageal and extra-esophageal symptoms (e.g. chronic cough).

In humans, pain is a multimodal experience composted of sensory, physiological and psychological aspects. In order to mimic the clinical situation, experimental models should be based on multimodal testing regimens in which different receptors and central nervous system mechanisms are activated.

Advances in esophageal sensory stimulation have established that both typical and atypical symptoms may not only arise from acid reflux, but also from reflux events with less acidic pH (pH 4-7). In GERD patients with symptoms that persist in spite of PPIs, ongoing weakly acidic reflux is now well established as the main underlying factor.

The basis for symptom generation during weakly-acidic reflux events remains to be determined, but acid sensitivity in the pH range 4-7, mechanical distention (enhanced by air in the refluxate), sensitivity to other chemical factors (e.g. bile) and esophageal hypersensitivity to physiological levels of reflux have all been proposed.

HYPOTHESIS The investigators speculated that visceral hypersensitivity plays an important role in symptom perception. This is suggested by the reflux parameters that are usual within the physiological number during PPI therapy.

Naloxone is indicated for the complete reversal of opioid depression, including respiratory depression, induced by natural and synthetic opioids. Naloxone is also indicated for diagnosis of suspected or known acute opiod overdosage. Off label it is also used for alcoholic coma, Alzheimer's disease, schizophrenia, opioid addiction and narcotic induced pruritis. Methylnaltrexone bromide (Relistor) is indicated for the treatment of opioid-induced constipation in patients with advanced illness who are receiving palliative care, when response to laxative therapy has not been sufficient.

AIM The aim of the study was to investigate the effect of naloxone (IV or IM administration) and methylnaltrexone (subcutaneous administration) on esophageal sensitivity, in a group of healthy volunteers in order to evaluate the role of endogenous opiods in symptom perception in gastro-esophageal reflux disease..

METHODS Studies were performed in 12 healthy volunteers, to have sufficient data to compare subjects mutual and to be able to make conclusions. Since this concerns measurements with drugs that were never tested in this field of work, the investigators did not have information regarding esophageal sensitivity after administration of these different substances. Because of previous experience with these types of measurements (i.c. multimodal stimulation with other substances), the investigators concluded that a number of 12 healthy volunteers was sufficient to detect a 30% difference with a 5% significance level.

For safety reasons, subjects were prohibited to drive a vehicle or work with heavy machinery on the day of the study. Each subject that was willing to participate was submitted to a physical examination. Medical history was taken and the use of medication was inquired.

Studies were performed using a multimodal esophageal stimulation probe which allows chemical, mechanical, electrical and thermal stimulations of the esophagus in one single protocol.

During each stimulation, subjects were instructed to record perception of symptoms using an electronic VAS meter. This device allows the subject to scale perception and pain on a scale from 0 to 10.

First perception (VAS=1), pain perception threshold (VAS=5) and pain tolerance threshold (VAS=7) were recorded. All types of esophageal stimulations were immediately terminated when the pain tolerance threshold was reached. At the time when the pain tolerance threshold was reached (VAS=7), the subjects were asked to draw the referred pain area, to identify where the pain was located.

Thermal stimulation Thermal stimulation was performed by re-circulating a saline solution (NaCl 0.09%), heated by a water bath, through the balloon mounted on the probe. Stimulation temperature was steadily increased by increasing the flow rate from the water bath to the balloon. Flow rate will be controlled by a computer operated pump. The volume in the balloon was kept constant at 5ml to avoid mechanical stimulation of the esophagus.

A temperature sensor present in the balloon montinuously monitored the stimulation temperature, which was displayed on a computer display throughout the study.

Mechanical stimulation Mechanical stimulation was performed by distention of the balloon mounted on the probe. The flow of saline (NaCl 0.09%) into the balloon, inducing the distention, was regulated by a computer controlled pump. The volume in the balloon was displayed on the computer screen throughout the stimulation. Mechanical stimulations were performed with water of 37°C, to avoid thermal stimulation of the esophagus.

Mechanical stimulation was preceded by a preconditioning period during which the balloon was distended until the pain perception threshold (VAS=5) was reached. This preconditioning period was used to precondition the esophageal tissue and to allow the subject to get used to the feeling of mechanical distention.

Electrical stimulation Electrical stimulation was performed by 2 stimulation electrodes mounted on proximal to the balloon. Electrical block pulses were given using a standard electrical stimulator. Single burst pulses were given with duration of 1ms at 200Hz. The amplitude of the pulses was steadily increased, with steps of 0.5mA and an interval of 15sec. The maximum intensity is limited to 60 mA, as previous studies have shown atrial capturing with higher intensities. ECG monitoring was performed as a safety measure during the electrical stimulations of the esophagus.

Chemical stimulation Chemical stimulation was performed in distal esophagus by infusing an acidic solution (HCl 0.1N) in the esophagus. Chemical stimulations were controlled by a peristaltic infusion pump with a flow rate of 2ml/min.

Naloxone/Methylnaltrexone or placebo administration As test solutions, naloxone (bolus of 0.4 mg followed by continuous infusion 20 µg/kg/h) or methylnaltrexone bromide (12 mg s.c., Relistor 0.6ml administrated subcutaneously) were administered. During placebo sessions, a physiological solution (saline 0.9%), was administered IV and SC. Over time, each participant received placebo or naloxone or methylnaltrexone bromide in the first session in a random sequence. In the second and third session, the subject received one of the other products that he/she did not receive the first time.

STUDY OUTLINE After an overnight fast subjects were expected at the endoscopy unit of the UZ Gasthuisberg, where the study was performed. Three sessions were scheduled for every subject: one placebo, one naloxone session and one methylnaltrexone session, with at least one week interval between each of them. Sessions were run in a double blind way, as far as the placebo or drugs are concerned. The order of placebo and drug administration was randomized by drawing cards from a box of cards determining the sequence.

The volunteer received placebo, naloxone or methylnaltrexone at the beginning of the session.

The multimodal stimulation probe was positioned through the mouth. After the probe was positioned in the esophagus, it was fixed to the chin and the subject remained in a bed, in semi-recumbent position for the entire study period. Esophageal stimulation was performed immediately after intubation.

Before the actual stimulations started, there was an adaptation period for the subjects, to get used to the feeling of the probe and to provide instructions for the correct use of the VAS meter since VAS scores were monitored during each type of stimulation.

All stimulations were immediately stopped at the moment the subject reached the pain tolerance threshold (VAS=7).

ANALYSIS Temperature, volume, and electrical current will be measured at VAS=1 (first perception), VAS=5 (pain perception threshold) and VAS=7 (pain tolerance threshold) and were used to determine esophageal sensitivity. Esophageal sensitivity for the four different stimuli (temperature, mechanical, electrical and chemical) were compared between the three conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* No history of gastrointestinal symptoms or complaints

Exclusion Criteria:

* A history of allergic reaction to naloxone or methylnaltrexone bromide or multiple allergies to several foods and drugs.
* Pregnancy, lactation.
* Concomitant administration of monomine oxidase inhibitors (MAOI), verapamil or diltiazem or medications affecting esophageal motility.
* Significant co-morbidities (neuromuscular, psychiatric, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic).
* Prior history of esophageal, Ear-Nose-Troat or gastric surgery or endoscopic anti-reflux procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Measurement of changes in esophageal sensitivity after IV naloxone or IM methylnaltrexone administration | 3 sessions per HV with at least one week interval, duration of each session: approximately 2 hours. Temperature stimulation: 30 minutes
  Investigation of the effect of Naloxone and methylnaltrexone-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the Temperature values (°C) of the stimulation tests between the placebo and naloxone and methylnaltrexone condition to see if CRH affects the sensitivity to increasing temperature
Measurement of changes in esophageal sensitivity after IV naloxone or IM methylnaltrexone administration | 3 sessions per HV with at least one week interval, duration of each session: approximately 2 hours. Mechanical stimulation: 30 minutes
  Investigation of the effect of Naloxone and methylnaltrexone-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the balloon volumes (volume in ml) of the stimulation tests between the placebo and Naloxone and methylnaltrexone condition to see if Naloxone and methylnaltrexone affect the sensitivity to increasing balloon volume.
Measurement of changes in esophageal sensitivity after IV naloxone or IM methylnaltrexone administration | 3 sessions per HV with at least one week interval, duration of each session: approximately 2 hours. Electrical stimulation: 30 minutes
  Investigation of the effect of Naloxone and methylnaltrexone-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the tolerated intensity of the electrical pulses (mA) of the stimulation tests between the placebo and Naloxone and methylnaltrexone condition to see if Naloxone and methylnaltrexone affect the sensitivity to increasing electrical pulses.
Measurement of changes in esophageal sensitivity after IV naloxone or IM methylnaltrexone administration | 3 sessions per HV with at least one week interval, duration of each session: approximately 2 hours. Chemical stimulation: 30 minutes
  Investigation of the effect of Naloxone and methylnaltrexone-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the volume of infused acid (ml) of the stimulation tests between the placebo and Naloxone and methylnaltrexone condition to see if Naloxone and methylnaltrexone affect the sensitivity to acid infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PhD, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: No